CLINICAL TRIAL: NCT00601471
Title: Effects of Proximal and Distal Tibiofibular Joint Manipulation on Lower Extremity Muscle Activation, Ankle Range of Motion, and Functional Outcome Scores in Individuals With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: American Physical Therapy Association (Other)
Responsible Party: Jay Kertel, PhD, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12966
Record Dates: First submitted 2008-01-14; First posted 2008-01-28 (Estimated); Last update posted 2010-06-24 (Estimated); Status verified 2010-06

CONDITIONS: Ankle Sprain; Ankle Injuries; Sprain
Keywords: ankle sprain; ankle injuries; sprains and strains
MeSH Terms: conditions — Ankle Injuries; Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): proximal tibiofibular manipulation
  Interventions: Other: proximal tibiofibular manipulation
- 2 (Experimental): distal tibiofibular manipulation
  Interventions: Other: distal tibiofibular manipulation
- 3 (No Intervention): no treatment
  Interventions: Other: no intervention

INTERVENTIONS:
Other: proximal tibiofibular manipulation — proximal tibiofibular manipulation
  Arms: 1
Other: distal tibiofibular manipulation — distal tibiofibular manipulation
  Arms: 2
Other: no intervention — no intervention / control
  Arms: 3

SUMMARY:
The overall aim of this project is to determine the effect of a tibiofibular joint manipulation on the neuromuscular response of the fibularis longus and soleus muscles in individuals with chronic ankle instability. Another aim of this study is to determine the long term effects of a tibiofibular joint manipulation on range of motion and self-reported function.

We hypothesize that a manipulation applied at the distal tibiofibular joint will result in greater muscle activation, improved functional dorsiflexion ROM, and increases in FAAM scores compared to a tibiofibular joint manipulation applied at the proximal joint. We further hypothesize that both distal and proximal tibiofibular joint manipulations will result in greater muscle activation, improved functional dorsiflexion ROM, and increases in FAAM scores than no treatment at all.

DETAILED DESCRIPTION:
Muscle weakness is a common impairment following injury to a joint. Individuals with lateral ankle sprains have been shown to demonstrate weakness and inhibition of the fibularis longus and soleus muscles. Recently, changes in the positional alignment of the talus, tibia, and fibula have been implicated in a subpopulation of individuals with chronic ankle instability (CAI). Clinically this manifests as a decrease in the posterior glide of the talus and decreased dorsiflexion ROM. Another positional fault has been noted to occur between the distal tibiofibular joint. A subpopulation of individuals with a history of CAI have demonstrated a slight anterior displacement of the fibula relative to the tibia. The cause of the malpositioning is unknown, but manual therapeutic interventions may offer the ability to restore normal joint arthrokinematics and muscle function. It is unknown if the correction of this positional fault will have an effect on muscle inhibition about the ankle.

Since muscle inhibition is a neurological reflexive reaction, it is thought that traditional strengthening treatment techniques may not fully address this dysfunction. Manual therapeutic interventions can have dual effects on the neuromuscular system and restore normal joint arthrokinematics. Evidence suggests a joint manipulation is able to disinhibit or even facilitate local and distant muscles. This likely occurs due to the afferent response from the structures in and around the manipulated joint. Comprehensive treatment interventions which restore normal joint function, optimal motoneuron pool excitability, strength, and pain-free previous level of function need to be developed to prevent future dysfunction and osteoarthritis.

Currently no study has examined the effects of tibiofibular joint manipulation on the neuromuscular response of ankle musculature or the effects on range of motion and function. The purpose of this study is to examine the acute effects of a tibiofibular joint manipulation on the neuromuscular response of the fibularis longus and soleus muscles and to determine the long term effects on range of motion and function in individuals with CAI.

The first research question will address how a tibiofibular joint manipulation immediately affects the activation of the fibularis longus and soleus muscles. The second question will address how this joint manipulation affects range of motion and functional outcomes over a three week period. Changes in ankle dorsiflexion range of motion (ROM), navicular drop, Step Down Test, Balance Error Scoring System, and the Foot and Ankle Ability Measure (FAAM) will be used to determine if clinically significant changes occurred during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* History of more than one ankle sprain
* unilateral or bilateral
* Complaint of chronic ankle instability (CAI) and qualified according to
* 4 "YES" responses on the Ankle Instability Instrument (AII)
* Scoring at least an 85 on the Foot and Ankle Ability Measure (FAAM)

Exclusion Criteria:

* Lower extremity injury in the past 6 months (including lateral ankle sprain)
* Currently receiving physical therapy for a lower extremity injury
* Have a previous history of lower extremity surgery
* Have diagnosed ankle osteoarthritis or rheumatoid arthritis
* Currently pregnant or breast feeding
* History of connective tissue disorders (like Marfan's Syndrome or Ehlers Danlos Disease)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2007-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Changes in muscle activation | over a three week period

SECONDARY OUTCOMES:
changes in functional range of motion | over a 3 week period
changes in function | over a three week period

CONTACTS AND LOCATIONS:
Overall Officials: Jay Hertel, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States